CLINICAL TRIAL: NCT06722781
Title: UpLift-X Trial 1: A Cluster Factorial Randomised Controlled Trial of Digitally-enabled Group Psychotherapy for Common Mental Disorders
Brief Title: Trial of an Online Group Psychotherapy Intervention for Common Mental Health Disorders
Acronym: UpLift-X
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rotherham Doncaster and South Humber NHS Foundation Trust (Other Government)
Collaborators: Innovate UK (Other Government); University of Sheffield (Other); MindLife UK Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: RDaSH0348
Record Dates: First submitted 2024-10-07; First posted 2024-12-09 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Common Mental Health Problems; Anxiety; Depression Disorders
Keywords: Psychological interventions; Internalizing disorders; High intensity CBT; Common mental health problems; Unified Protocol; Digitally-enabled therapy; Group therapy; Digital Health Technology; NHS Talking Therapies; Personalised treatment; Pragmatic clinical trial; Transdiagnostic
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Pragmatic factorial cluster randomised controlled trial of a transdiagnostic treatment for common mental health problems
Masking Description: The cluster randomisation sequence will be generated by a research assistant who is not involved in recruitment, treatment delivery or data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Standard Unified Protocol (UP) (Active Comparator): Standard sequence of UP modules, 1, 2, 3, 4, 5 6, 7, 8.
  Interventions: Behavioral: Unified Protocol
- UP Sequence 1 (Active Comparator): Sequence of modules, 1, 2, 5, 7, 4, 3, 6, 8.
  Interventions: Behavioral: Unified Protocol
- UP Sequence 2 (Active Comparator): Sequence of modules, 1, 2, 6, 3, 5, 7, 8.
  Interventions: Behavioral: Unified Protocol
- UP Sequence 3 (Active Comparator): Sequence of modules, 1, 2,4, 6, 7, 5, 3, 8.
  Interventions: Behavioral: Unified Protocol
- UP Sequence 4 (Active Comparator): Sequence of modules, 1, 2, 7, 5, 3, 4, 6, 8.
  Interventions: Behavioral: Unified Protocol

INTERVENTIONS:
Behavioral: Unified Protocol — The UP is a transdiagnostic treatment that was designed to be relevant to a wide range of emotional disorders, given the common co-occurrence of depression, anxiety, somatoform and dissociative symptoms. It is based on Cognitive and Behavioural Therapy (CBT) and emotion regulation theories, and the aim is to support patients to apply a series of emotion regulation skills that target the core common vulnerabilities that underlie a range of mental health problems: neuroticism, low perceived control, and overestimation of threat. Contents are organised across 8 modules delivered online across 12 weekly 1.5 hour sessions and will include a combination of internet-based resources (self-monitoring questionnaires, psychoeducational videos, skills practices linked to each module) and group therapy sessions delivered by a qualified cognitive behavioural therapist.
  Other Names: Transdiagnostic UP; Barlow's Unified Protocol for emotional disorders

SUMMARY:
The goal of this clinical trial is to understand how to deliver online group therapy for adults with common mental health problems in a personalised way. This study will test a new online group therapy program for various common mental health problems like anxiety and depression. The therapy is based on an approach called the Unified Protocol, which includes eight modules teaching different coping skills. The therapy will be delivered via a video call and a website, which will also have helpful videos and information about coping skills.

Aims:

1. Does changing the order of the therapy modules affect how well treatment works or how many patients drop-out of treatment?
2. Do some modules work better for different patients based on their individual features and if patients receive the therapy module that is most likely to be helpful for them first, does it mean they have a better chance of feeling better by the end of treatment?
3. Does online group therapy work as well to treat common mental health problems as standard care (individual cognitive behavioural therapy [CBT])?

Hypotheses:

1. Changing the order of therapy modules will not change how well therapy works or how many people drop-out.
2. Patients with specific profiles (based on their individual characteristics) will benefit more from some treatment modules and will see greater improvements in their symptoms if they received their best therapy module before other modules
3. There will be no differences in overall treatment outcome or dropout rates when comparing online group therapy vs. individual CBT

Researchers will compare whether delivering the modules in different orders, with five different versions of the treatment, to see if changing the order of therapy modules affects how well it works or drop-out rates. Researchers will test how best to match patients to the most helpful parts of treatment for them. The group therapy outcomes and costs will also be compared to data from patients who have had individual CBT to see how the intervention compares to standard care.

Participants will:

* Complete online symptom questionnaires before treatment starts and before each therapy session
* Attend 12 weekly group therapy sessions delivered by a video call on a website (called Uplift-X).
* Access online resources like videos and practice exercises to use between therapy sessions.
* Complete the online symptom questionnaires again at the end of treatment and 6 months later.

DETAILED DESCRIPTION:
The study protocol - including a full statistical analysis plan was pre-registered and made publicly accessible in the Open Science Framework on the 4th of October 2024 (available here - https://osf.io/vup9c/).

A pragmatic, multi-site, cluster factorial randomised controlled trial, involving National Health Service (NHS) Talking Therapies (NHS-TT) services for anxiety and depression (formerly known as IAPT services) in England. The "UPLift" digitally enabled group intervention, based on the Unified Protocol, will be available to patients with common mental disorders (and comorbidities) that are eligible to receive high intensity Cognitive Behavioural Therapy (CBT) in NHS-TT services, following national guidelines (National Collaborating Centre for Mental Health, 2024). The Unified Protocol is a transdiagnostic treatment that was designed to be relevant to a wide range of emotional disorders, given the common co-occurrence of depression, anxiety, somatoform and dissociative symptoms. It is based on CBT and emotion regulation theories, and aims to support patients to apply a series of emotion regulation skills that target the core common vulnerabilities that underlie a range of mental health problems: neuroticism, low perceived control, and overestimation of threat. The protocol follows the principle of parsimony, by including the minimum number of empirically validated techniques that would make it accessible, uncomplicated, and effective for the maximum number of patients with various combinations of symptoms and problems. Contents are organised across 8 modules delivered online at 12 weekly 1.5 hour sessions and will include a combination of internet-based resources (self-monitoring questionnaires, psychoeducational videos, skills practices linked to each module) and group therapy sessions delivered by a qualified cognitive behavioural therapist.

The unit of randomisation (cluster) will be each participating NHS-TT service. NHS Trusts are wider organisations that manage one or more NHS-TT services, so the unit of randomisation is the local team. All patients treated in the same local area service will be members of the same cluster. Participating services will be randomly allocated to one of 5 arms. Each arm will include the same 12-session online group Unified Protocol treatment but organised in a different sequence. The first two modules will remain fixed at the start of the intervention, as these introduction sessions are necessary to orient all patients to the treatment and to establish a cohesive group process. Similarly, the final module is fixed at the end of the intervention, as it includes an overall review of all coping skills, and it focuses on relapse prevention. The middle modules cover specific emotion regulation skills and are most amenable to personalisation (e.g., some may be more or less effective for specific patients). These prescriptive modules will be delivered in different sequences across each of the trial arms.

Participants will complete baseline measures on entry to the study, weekly symptom outcome measures prior to each session and a post-treatment (session 12) and 6-month follow-up survey. The primary outcome will be Negative affectivity (NA), based on a composite score pooling items from Patient Health Questionnaire-9 (PHQ-9; depression), Generalized Anxiety Disorder-7 scale (GAD-7; anxiety) and Work and Social Adjustment Scale (WSAS; functioning). Secondary outcomes will be Quality of life (EuroQol - 5 dimensions; EQ5D), Wellbeing (Warwick and Edinburgh Mental Wellbeing Scale; WEMWBS) and drop out from treatment.

Researchers will also collect anonymised clinical health records for all patients accessing individually delivered CBT in the participating services during the period of the clinical trial. These data will include demographics, clinical care and clinical outcomes. This will enable researchers to undertake comparisons of clinical and cost-effectiveness using a case-control matching strategy described in the statistical analysis plan.

The statistical analysis plan will be carried out in three stages linked to each of the objectives of the study.

Objective 1: compare outcomes of different UP module sequences This will be the primary analysis, based on which the sample size calculation is based. Cases with missing post treatment (12th session) data-points in the dependent variable will be imputed using the MissForest R package using all baseline variables as predictors. Imputations will be carried out separately for each trial arm. The analysis will apply a linear multilevel (mixed effects) model, where patients will be nested within groups, entering a random effect for the group-level. The dependent variable will be the post-treatment Negative Affectivity (NA) score, entering trial arm as an independent variable, controlling for baseline NA. Models will be developed in sequential steps and model fit indices (AIC, BIC, -2LL) will be examined after each modelling step. Researchers will retain and interpret the best-fitting and most parsimonious model achieved through this stepwise process, using the -2 loglikelihood ratio test to compare models. The intra-cluster correlation coefficient (ICC) will be reported as an index of variability in treatment outcomes attributable to the group-level. Between-group effect sizes (Cohen's d) will be calculated and reported for each contrast (e.g., standard UP sequence vs. other sequences).

Secondary analysis: The above analysis plan will be repeated using a logistic multilevel model with dropout as the dependent variable. The dropout variable will be derived from group therapy attendance records, where cases that attended more than half (≥6) sessions will be grouped into the reference category (code = 0) and cases that attended less than half (≤5) will be classed as cases that dropped out (code = 1).

Objective 2: develop a personalised module selection method Cases with missing data-points in the dependent variable will be imputed using the MissForest R package using all baseline variables as predictors, with separate imputations in the training/validation partitions, and within each trial arm. Reliable improvement (RI) refers to a reduction in symptom severity in between two time-points, which is greater in magnitude than the reliable change index for the psychometric measure. Following this definition, the investigators will class cases using a binary variable denoting whether they did (code = 1) or did not (code = 0) have reliable improvement after exposure to a prescriptive Unified Protocol module. This coding will enable us to identify cases that experience reliable symptomatic improvements after exposure to each of the target modules, regardless of where the module is located (e.g., towards the start, middle or end of the intervention) in the group intervention they have been allocated to. This methodology will enable researchers to control for sequencing and early response effects, to identify the profile of patients who have a favourable response to each specific module.

Sample partitioning: The full trial sample will be randomly partitioned into training and validation subsets using a 60:40 split, with a balanced number from each of the 5 trial arms in each training-partition split. This will ensure that 396 cases will be randomly selected into the training partition, exceeding the minimum sample size of 300 necessary to train a reliable clinical prediction model using supervised machine learning.

Model development and optimisation (in the training partition): Researchers will produce a total of 5 machine learning prediction models, one for each prescriptive UP module. Each trained model will process inputs (patients' baseline features) and will output [a] a predicted classification and [b] a corresponding predicted probability pertaining to the classification. The logic of these algorithms is to answer the following question: Given these patient characteristics, how likely is it that this specific patient will experience reliable improvement after accessing module X? Cross-validation strategy (in the validation sample): The statistical accuracy and clinical utility of the machine learning models will be evaluated in the validation strategy by comparing the algorithm predictions against the observed outcomes and comparing outcomes for patients who received their optimal module first compared to patients who did not.

Secondary analysis: The above machine learning analysis and cross-validation strategy will be repeated to train a binary classifier with dropout as the dependent variable. The dropout variable will be derived from group therapy attendance records, where cases that attended more than half (≥6) sessions will be grouped into the reference category (code = 0) and cases that attended less than half (≤5) will be classed as cases that dropped out (code = 1).

Objective 3: evaluate the effectiveness of digitally enabled UP group therapy vs. individual CBT This analysis will include [a] a subgroup of clinical trial participants who were randomly assigned to the arm where the UP protocol was delivered in the standard sequence, and [b] a matched sample of patients who accessed individual high intensity CBT in the participating NHS-TT services. The data for the individual CBT cases will be sampled from electronic health records. CBT cases that meet the trial inclusion criteria listed will be selected for this analysis, only including cases where the primary presenting problem is identifiable in clinical records and where baseline severity scores (PHQ-9, GAD-7, WSAS) are available at their first attended CBT session. Cases with missing post-treatment (last attended session) data-points in the dependent variable will be imputed using the MissForest R package using all covariates as predictors. Imputations will be carried out separately for each group (individual CBT; standard UP group therapy). Post-treatment clinical outcomes (NA scores) will be compared between cases accessing the standard group UP protocol versus individual CBT cases using doubly robust estimation, which combines an adjustment for non-random allocation to treatments, and a covariate-adjusted regression model to test the causal effect of exposure to an intervention.

Secondary analyses: The above analysis will be repeated to compare outcomes using disorder-specific measures (PHQ-9, GAD-7, ADSM) for cases with the relevant diagnoses. Between-group effect sizes (Cohen's d) will be calculated and reported for each comparison.

Health economic analysis: An economic analysis will be conducted from the NHS and Personal Social Services perspective. A cost-utility analysis will use quality-adjusted life years (QALYs derived from the EQ-5D questionnaire, and tariff based on the UK public value set) as the measure of quality of life, using post-treatment (last-attended session) data on the NA scale in the primary analysis, and 3-month follow-up data in a secondary analysis. Health and social services resource use will be valued using NHS reference costs and the personal and social services resource use database (PSSRU). Investigators will estimate the incremental cost effectiveness ratio for group therapy versus individual CBT, using bootstrapping to estimate confidence intervals. Decision uncertainty will be presented on a cost-effectiveness acceptability curve. Additional sensitivity analyses will be conducted for resource use and unit costs. A sensitivity analysis will control for baseline costs. Scenario analyses will explore alternative costing perspectives; that is, NHS and NHS/PSS perspectives. Results of the cost-effectiveness analysis will be reported in line with the Consolidated Health Economic Evaluation Reporting Standards 2022 Statement.

ELIGIBILITY:
Inclusion Criteria:

* 17 years old and over
* Literate and fluent in the English language, which would enable group interactions and learning via online materials
* With access to an internet-connected device (e.g., computer, phone) and confidential space
* Referred to NHS-TT services
* Assessed by a qualified psychological professional and deemed to be eligible for high intensity CBT (this includes low risk of harm to self or others)
* Currently on waiting list for high intensity CBT and not accessing any other psychological interventions. This includes patients accessing pharmacotherapy but who are additionally seeking psychological treatment
* Presenting symptoms of one or more internalizing disorders (major depressive disorder, generalised anxiety disorder, panic disorder, agoraphobia, specific phobias, somatoform disorder, obsessive-compulsive and related disorders, body dysmorphic disorder, post-traumatic stress and related disorders)

Exclusion Criteria:

* 16 years old and under
* Not able to speak or read English fluently, which would require more individualised support with interpreters
* No access to internet-connected device or confidential space to engage with digital intervention
* Not involved with NHS-TT services
* Assessed by a qualified psychological professional and not deemed to be eligible for high intensity CBT on the basis of mental health condition and/or risk assessment (e.g., acute risk of suicide at the time of assessment)
* Already accessing a high intensity psychotherapy or other forms of psychological treatment (e.g., private therapy, counselling)
* Presenting with symptoms of eating disorders, substance use disorders, psychotic disorders, personality disorders, bipolar disorders identified at the time of initial assessment.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Post-treatment Negative Affectivity (NA) scale | Through study completion, an average of 11 months
  A transdiagnostic construct that includes commonly occurring symptoms of low mood, negative thoughts, fear/anxiety, social and interpersonal difficulties. NA can be measured by pooling all items from the PHQ-9, GAD-7 and WSAS into a single scale which attributes specific weights to each item according to their strength of association with an underlying dimension of general psychological distress. To derive this NA scale, we will apply the item-weighting methodology proposed by. This involves multiplying the raw item scores across all three questionnaires with the non-standardized factor loadings. This yields a continuous NA severity score ranging between 0 and 69.58, with a reliable change index.

SECONDARY OUTCOMES:
Quality of Life (EuroQol - 5 dimensions; EQ5D) | Through study completion, an average of 11 months
  The EuroQol Group 5-Dimension self-report questionnaire (EQ-5D) measures health-related quality of life across five domains: mobility, self-care, daily activities, pain/discomfort, and depression/anxiety. This measures yields a continuous score with a range between -0.446 to 1.00, where higher scores indicate better quality of life.
Wellbeing (Short-form Warwick and Edinburgh Mental Wellbeing Scale; SWEMWBS) | Through study completion, an average of 11 months
  The Short-form Warwick and Edinburgh Mental Wellbeing Scale (SWEMWBS) is a 7-item self-report scale that measures psychological well-being, with a continuous score ranging between 7 and 35, where a higher score indicates better well-being.
Therapy drop-out | 12 weeks (at the end of therapy).
  The dropout variable will be derived from group therapy attendance records, where cases that attended more than half (≥6) sessions will be grouped into the reference category (code = 0) and cases that attended less than half (≤5) will be classed as cases that dropped out (code = 1).

OTHER OUTCOMES:
Healthcare service utilisation (Modified Adult Service Use Schedule; AD-SUS) | Through study completion, an average of 11 months
  A modfied measure of healthcare service utilisation for health economic analysis. The measure captures binary (yes/no) information about which healthcare services participants have used in the last 3 months and how many times. There is no minimum or maximum score. The responses provided are combined with known healthcare cost values to conduct economic analyses of the study intervention and subsequent impact on other healthcare usage.
Group alliance (Group Climate Questionnaire-Short; GCQ-S) | 3 Weeks (Session 3)
  To control for group alliance levels, participants will complete the 12-item Group Climate Questionnaire-Short (GCQ-S). There are 3 scales; Enaged (scored 0-30 where higher scores show better engagement), Conflict (scored 0-24 where higher scores show greater conflict), and Avoiding (scored 0-18 where higher scores show more avoidance).

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Delgadillo, PhD, Principal Investigator — University of Sheffield
Locations (2):
- United Kingdom (2):
  - Rotherham Doncaster and South Humber NHS Foundation Trust, Doncaster, South Yorkshire
  - Devon Partnership NHS Trust, Exeter

IPD SHARING:
Plan to Share IPD: No
The study dataset will be only accessible to collaborators named in this study protocol, in a fully pseudonymised format. Study data will not be made available in a publicly accessible repository. Requests for data access are to be made in writing to the Chief Investigator, and will only be granted to qualified academic researchers who provide a study protocol and after this protocol has been pre-registered in a public repository such as the open science framework.

REFERENCES:
- [Background] Howard KI, Lueger RJ, Maling MS, Martinovich Z. A phase model of psychotherapy outcome: causal mediation of change. J Consult Clin Psychol. 1993 Aug;61(4):678-85. doi: 10.1037//0022-006x.61.4.678. PMID 8370864
- [Background] Fisher AJ, Bosley HG, Fernandez KC, Reeves JW, Soyster PD, Diamond AE, Barkin J. Open trial of a personalized modular treatment for mood and anxiety. Behav Res Ther. 2019 May;116:69-79. doi: 10.1016/j.brat.2019.01.010. Epub 2019 Feb 21. PMID 30831478
- [Background] Emsley, R., Lunt, M., Pickles, A., & Dunn, G. (2008). Implementing double-robust estimators of causal effects. The Stata Journal, 8(3), 334-353. https://doi.org/10.1177/1536867X0800800302
- [Background] Dolan N, Simmonds-Buckley M, Kellett S, Siddell E, Delgadillo J. Effectiveness of stress control large group psychoeducation for anxiety and depression: Systematic review and meta-analysis. Br J Clin Psychol. 2021 Sep;60(3):375-399. doi: 10.1111/bjc.12288. Epub 2021 Apr 6. PMID 33822376
- [Background] Delgadillo J, Kellett S, Ali S, McMillan D, Barkham M, Saxon D, Donohoe G, Stonebank H, Mullaney S, Eschoe P, Thwaites R, Lucock M. A multi-service practice research network study of large group psychoeducational cognitive behavioural therapy. Behav Res Ther. 2016 Dec;87:155-161. doi: 10.1016/j.brat.2016.09.010. Epub 2016 Sep 20. PMID 27685938
- [Background] Briggs AH, Wonderling DE, Mooney CZ. Pulling cost-effectiveness analysis up by its bootstraps: a non-parametric approach to confidence interval estimation. Health Econ. 1997 Jul-Aug;6(4):327-40. doi: 10.1002/(sici)1099-1050(199707)6:43.0.co;2-w. PMID 9285227
- [Background] Ayuso-Bartol, A., Gómez-Martínez, M. Á., Riesco-Matías, P., Yela-Bernabé, J. R., Crego, A., & Buz, J. (2024). Systematic review and meta-analysis of the efficacy and effectiveness of the unified protocol for emotional disorders in group format for adults. International Journal of Mental Health and Addiction. Advance online publication. https://doi.org/10.1007/s11469-024-01330-z
- [Background] Barkowski S, Schwartze D, Strauss B, Burlingame GM, Barth J, Rosendahl J. Efficacy of group psychotherapy for social anxiety disorder: A meta-analysis of randomized-controlled trials. J Anxiety Disord. 2016 Apr;39:44-64. doi: 10.1016/j.janxdis.2016.02.005. Epub 2016 Feb 10. PMID 26953823
- [Background] Beard JIL, Delgadillo J. Early response to psychological therapy as a predictor of depression and anxiety treatment outcomes: A systematic review and meta-analysis. Depress Anxiety. 2019 Sep;36(9):866-878. doi: 10.1002/da.22931. Epub 2019 Jun 24. PMID 31233263
- [Background] Bohnke JR, Lutz W, Delgadillo J. Negative affectivity as a transdiagnostic factor in patients with common mental disorders. J Affect Disord. 2014 Sep;166:270-8. doi: 10.1016/j.jad.2014.05.023. Epub 2014 May 27. PMID 25012441
- [Background] Cassiello-Robbins C, Southward MW, Tirpak JW, Sauer-Zavala S. A systematic review of Unified Protocol applications with adult populations: Facilitating widespread dissemination via adaptability. Clin Psychol Rev. 2020 Jun;78:101852. doi: 10.1016/j.cpr.2020.101852. Epub 2020 Apr 20. PMID 32360953
- [Background] Funk MJ, Westreich D, Wiesen C, Sturmer T, Brookhart MA, Davidian M. Doubly robust estimation of causal effects. Am J Epidemiol. 2011 Apr 1;173(7):761-7. doi: 10.1093/aje/kwq439. Epub 2011 Mar 8. PMID 21385832
- [Background] Karyotaki E, Riper H, Twisk J, Hoogendoorn A, Kleiboer A, Mira A, Mackinnon A, Meyer B, Botella C, Littlewood E, Andersson G, Christensen H, Klein JP, Schroder J, Breton-Lopez J, Scheider J, Griffiths K, Farrer L, Huibers MJ, Phillips R, Gilbody S, Moritz S, Berger T, Pop V, Spek V, Cuijpers P. Efficacy of Self-guided Internet-Based Cognitive Behavioral Therapy in the Treatment of Depressive Symptoms: A Meta-analysis of Individual Participant Data. JAMA Psychiatry. 2017 Apr 1;74(4):351-359. doi: 10.1001/jamapsychiatry.2017.0044. PMID 28241179
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Nahum-Shani I, Dziak JJ, Collins LM. Multilevel factorial designs with experiment-induced clustering. Psychol Methods. 2018 Sep;23(3):458-479. doi: 10.1037/met0000128. Epub 2017 Apr 6. PMID 28383950
- [Background] Sauer-Zavala S, Cassiello-Robbins C, Conklin LR, Bullis JR, Thompson-Hollands J, Kennedy KA. Isolating the Unique Effects of the Unified Protocol Treatment Modules Using Single Case Experimental Design. Behav Modif. 2017 Mar;41(2):286-307. doi: 10.1177/0145445516673827. Epub 2016 Oct 22. PMID 28198196
- [Background] Sauer-Zavala S, Cassiello-Robbins C, Ametaj AA, Wilner JG, Pagan D. Transdiagnostic Treatment Personalization: The Feasibility of Ordering Unified Protocol Modules According to Patient Strengths and Weaknesses. Behav Modif. 2019 Jul;43(4):518-543. doi: 10.1177/0145445518774914. Epub 2018 May 10. PMID 29742904
- [Background] Sauer-Zavala S, Southward MW, Stumpp NE, Semcho SA, Hood CO, Garlock A, Urs A. A SMART approach to personalized care: preliminary data on how to select and sequence skills in transdiagnostic CBT. Cogn Behav Ther. 2022 Nov;51(6):435-455. doi: 10.1080/16506073.2022.2053571. Epub 2022 Apr 27. PMID 35475947
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Stekhoven DJ, Buhlmann P. MissForest--non-parametric missing value imputation for mixed-type data. Bioinformatics. 2012 Jan 1;28(1):112-8. doi: 10.1093/bioinformatics/btr597. Epub 2011 Oct 28. PMID 22039212
- [Background] Tennant R, Hiller L, Fishwick R, Platt S, Joseph S, Weich S, Parkinson J, Secker J, Stewart-Brown S. The Warwick-Edinburgh Mental Well-being Scale (WEMWBS): development and UK validation. Health Qual Life Outcomes. 2007 Nov 27;5:63. doi: 10.1186/1477-7525-5-63. PMID 18042300
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- See also: Open Science Framework (OSF) pre-registration of research project including copy of full protocol and analysis plan. — https://osf.io/vup9c/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT06722781/Prot_SAP_000.pdf